CLINICAL TRIAL: NCT04114318
Title: The Role of Cycling-cognitive Dual-task Training in Early Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201600213A3
Record Dates: First submitted 2019-08-26; First posted 2019-10-03 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-08

CONDITIONS: Safety and Effectiveness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive-Cycling (Experimental): Dual-task cognitive-cycling training; cognitive and cycling training simultaneously
  Interventions: Other: Dual-task cognitive-cycling training
- Cycling (Active Comparator): Single-task cycling training; stationary bicycle exercise training
  Interventions: Other: Dual-task cognitive-cycling training

INTERVENTIONS:
Other: Dual-task cognitive-cycling training — Cognitive and cycling training simultaneously for dual-task cognitive-cycling training; stationary bicycle exercise training for single-task cycling training
  Other Names: Single-task cycling training

SUMMARY:
The purpose of the study will investigate the safety and effectiveness with eight-week cycling-cognitive dual-task training for early Parkinson's disease.

DETAILED DESCRIPTION:
Background: Parkinson's disease is a neurodegenerative disorder of the basal ganglia in which the production of dopamine is reduced, leading to the motor and non-motor impairment and the loss of automaticity. Recently, the results across studies have indicated that motor-cognitive dual-task deficits in individuals with neurologic disorders appear to be amenable to training. Improvement of dual-task ability in individuals with neurologic disorders holds potential for improving gait, balance, and cognition. The most recent European guideline provides a more graded view, stating that in Hoehn and Yahr stages 2 and 3 dual-task training may be safe and effective. An overview of current ongoing randomized controlled trials focusing on dual-task rehabilitation, gait training or treadmill training was the major motor-task. However, cycling augmented by cognitive training has not been evaluated. In addition, antioxidant capacity is unclear for Parkinson's disease patients with long-term, regular cycling training.

Study purpose: The purpose of the study will investigate the safety and effectiveness with eight-week cycling-cognitive dual-task training for early Parkinson's disease. The antioxidant capacity will be assessed as well.

Methods: Parkinson's disease patients will be assigned to cycling training, cycling-cognitive dual task training, and following 8 weeks. All of the subjects will complete 3 assessments at pre-training, post-4 weeks, and post-8 weeks. The outcome measures are clinical severity and disability, performance of gait-cognitive and cycling-cognitive, cognitive-task performance, peripheral-blood oxidative stress, adverse events, etc.

Significance: In this study, evidence-based practice as the foundation, and perspective to design a safe and effective cycling-cognitive dual-task training for early Parkinson's disease. It can be verified in the clinical application of these experiments feasibility (practice-based evidence).

ELIGIBILITY:
Inclusion Criteria:

* patients with Idiopathic Parkinson's disease (IPD)
* an age between 45 to 70 years
* asymmetrical onset of at least 2 of 3 cardinal sign
* Modified Hoehn and Yahr staging from 1 to 2.5 during off state
* Montreal cognitive assessment score of 26 or greater

Exclusion Criteria: The patients were ineligible if they had

* a neurological history other than Parkinson's disease
* ever undergone neurosurgery for Parkinson's disease
* had moderate to severe dyskinesia
* been unstable with medical or psychiatric co-morbidities, orthopedic conditions restricting exercise
* done more than 20 min of aerobic exercise over 3 sessions per week on their own

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Unified Parkinson's disease rating scale | 30 minutes
  There are 4 parts subscores: part 1 (0-16), part 2 (0-52), part 3 (0-96), part 4 (0-23). Total scale range 0-187 (summed part 1, 2, 3, 4), higher values represent a worse outcome.
Gait speed in cm/second | 5 minutes
  using GAITRite with a 3.66-meter long and 0.9-meter wide instrumented walkway
Step length in cm | 5 minutes
  using GAITRite with a 3.66-meter long and 0.9-meter wide instrumented walkway
Step width in cm | 5 minutes
  using GAITRite with a 3.66-meter long and 0.9-meter wide instrumented walkway
Step time in second | 5 minutes
  using GAITRite with a 3.66-meter long and 0.9-meter wide instrumented walkway
Double limb support time in second | 5 minutes
  using GAITRite with a 3.66-meter long and 0.9-meter wide instrumented walkway
Modified Hoehn and Yahr staging | 5 minutes
  scale range 0-5. The scale was originally described in 1967 and included stages 1 through 5. It has since been modified with the addition of stages 1.5 and 2.5 to account for the intermediate course of Parkinson disease.
Time up and go test in second | 2 minutes
  The Timed Up and Go test (TUG) is a simple test used to assess a person's mobility

SECONDARY OUTCOMES:
Cognitive performance | 10 minutes
  The cognitive performance was described as a composite score (%) = accuracy (%)/reaction time (ms) *100
Dual-task interference | 10 minutes
  The effect of the dual-task was calculated as the difference between single-task and dual-task performance expressed as a percentage of single-task performance
Adverse event | 5 minutes
  any complain from study subject

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Song Lu, MD, Principal Investigator — Chang Gung Memorial Hospital

IPD SHARING:
Plan to Share IPD: No
after publishing, we will share IPD

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-21): https://cdn.clinicaltrials.gov/large-docs/18/NCT04114318/Prot_SAP_000.pdf